CLINICAL TRIAL: NCT02726139
Title: Improved Factor VIII Inhibitor Evaluation
Acronym: IFIE
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Shire (Industry); Emory University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: BVARI_GG_2016_1
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2016-03

CONDITIONS: Hemophilia; Hemophilia A
Keywords: Factor VIII; inhibitor; assay
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — frozen plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emory University: Samples obtained at and shipped from Emory University
- University of Michigan: Samples obtained at and shipped from University of Michigan

SUMMARY:
Commercial one and two-stage factor VIII assays may not detect some clinically significant inhibitor antibodies. The purpose of the proposed study is to standardize and validate a platelet-based factor VIII activity assay with greater sensitivity to clinically important inhibitory antibodies. Investigators will evaluate the platelet-dependent inhibitory activity vs. conventional inhibitory activity in stored patient plasmas and correlate to bleeding histories

DETAILED DESCRIPTION:
Factor VIII activity assays are used to diagnose hemophilia A, to monitor treatment of these patients, to determine when inhibitory antibodies against factor VIII have developed, and to evaluate the activity of engineered pharmaceutical factor VIII products. Factor VIII activity has been measured with one and two-stage assays for more than fifty years. However, all existing assays have major shortcomings that are recognized by the FDA, the International Society for Thrombosis and Haemostasis, and pharmaceutical companies. The major deficiencies that have been identified are: 1) Factor VIII activity levels do not predict the risk of bleeding in patients with inhibitory antibodies. The degree of inhibition in these assays is less than required to explain patient bleeding. 2) The assays are only accurate over a range of 1 - 100% of normal factor VIII activity, while values of 0.1 - 1% are also clinically important. 3) The different approved assays give discrepant values for recombinant pharmaceutical factor VIII products, with a range of 2-fold difference between assays. This can lead to clinically important differences in dosing of factor VIII products from one region to another with corresponding risk of thrombosis or bleeding.

The preliminary data identify an additional deficiency of commercial assays that has not been anticipated. Commercial one and two-stage assays may not detect some clinically significant inhibitor antibodies. Thus, the purpose of the proposed studies is to standardize and validate a platelet-based factor VIII activity assay with greater sensitivity to clinically important inhibitory antibodies.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia A
* presence of inhibitory antibodies

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A and inhibitory antibodies that have agreed to store plasma and prospectively consented to testing to evaluate bleeding mechanism
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Bleeding exceeds risk predicted by factor VIII assay | 1 year
  annual bleeding rate exceeds the rate predicted from the residual factor VIII activity
Bleeding is in accord with the risk assigned by platelet-dependent factor VIII activity | 1 year
  annual bleeding rate is within the predicted range from residual factor VIII activity

CONTACTS AND LOCATIONS:
Locations (1):
- Boston VA Research Institute (BVARI), Boston, Massachusetts, United States